CLINICAL TRIAL: NCT06042192
Title: Open Label Trial to Evaluate the Adhesion of TK-254RX in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teikoku Seiyaku Co., Ltd. (Industry)
Collaborators: ClinSearch (Other); SocraTec R&D GmbH (Other); SocraMetrics GmbH (Industry); CRM Biometrics GmbH (Industry); Clinigen Clinical Supplies Management GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TK-254RX-0106
Record Dates: First submitted 2023-09-10; First posted 2023-09-18 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TK-254RX applied to Lower Arm, Lower thigh or Ankle (Experimental): For Group1, TK-254RX will be applied to left and right side (total of two TK-254RX per day) of the following predetermined application site by subjects.
  Day1: Lower Arm, Day2: Lower thigh, Day3: Ankle
  Interventions: Drug: TK-254RX
- TK-254RX applied to Upper Arm, Upper thigh or Lower leg (Experimental): For Group2, TK-254RX will be applied to left and right side (total of two TK-254RX per day) of the following predetermined application site by subjects.
  Day1: Upper Arm, Day2: Upper thigh, Day3: Lower leg
  Interventions: Drug: TK-254RX

INTERVENTIONS:
Drug: TK-254RX — Two TK-254RX per day to predetermined application site

SUMMARY:
This study is a multi center, multiple dose, open label trial to evaluate the adhesion of TK-254RX in healthy volunteers. The primary purpose of this study is to evaluate the adhesion of TK-254RX. Secondary purpose is to show TK-254RX is safe and to explore and compare adhesion assessment methods.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 to 64 years
* good state of health
* non-smoker or ex-smoker for at least 3 months
* written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the subjects participating in the clinical trial

Exclusion Criteria:

The following must not apply:

* any injury of body which may induce the restriction of body movement
* excessively hairy skin at application site
* current skin disorder or shaving hair at application site
* history of excessive sweating/hyperhidrosis inclusive of application site
* participation in a clinical study within 30 days before inclusion in the study or concomitantly
* drug or alcohol abuse in the opinion of the investigator
* pregnant and lactating women
* women of child-bearing potential who do not agree to apply highly effective contraceptive methods
* known hypersensitivity to active ingredient, its racemate or one of the excipients of the TK-254RX
* existing cardiac and/or haematological diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient
* existing hepatic and/or renal diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient
* known liver or kidney insufficiency
* existing gastrointestinal diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient
* history of relevant CNS and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
* systolic blood pressure < 90 or > 139 mmHg
* diastolic blood pressure < 60 or > 89 mmHg
* pulse rate < 50 bpm or > 90 bpm
* subjects who use any impermissible medication

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Characterization of adhesion 5 minutes prior to removal by the adhesion assessment by site staff with EFTS marked by site staff | 5 minutes prior to removal,
  Assessment/estimation by site staff with marked TK-254RX by site staff: A listing of individual values of percentage will be presented per time point and subject.
  Descriptive statistics (Number, arithmetic mean, standard deviation, median, minimum and maximum) will be presented per time point for adhesion marker assessment by site staff with marked TK-254RX by site staff (percentage values).

SECONDARY OUTCOMES:
Characterization of adhesion by visual estimation of subjects | before bedtime (-1hour), after waking up (+1hour), 5minutes prior to removal
  Visual Assessment by subjects with a 5 point-scale: A listing of classification (≥90%, ≥75% to <90%, ≥50% to <75%, >0% to <50%, completely detached) of adhesion per time point and subject will be given.
Characterization of adhesion by the adhesion assessment by site staff with EFTS marked by subjects | before bedtime (-1hour), after waking up (+1hour), 5minutes prior to removal
  Assessment/estimation by site staff with marked TK-254RX by subject:
  A listing of individual values of percentage will be presented per time point and subject.
  Descriptive statistics (Number, arithmetic mean, standard deviation, median, minimum and maximum) will be presented per time point for adhesion marker assessment by site staff with marked TK-254RX by subject (percentage values).
Comparison of the adhesion assessments between subjects and study staff | 5minutes prior to removal
  Three different adhesion assessments at 24hours as below will be performed. i. Visual assessment scale by subject ii. Assessment scale by site staff with marked TK-254RX by subject iii. Assessment scale by site staff with marked TK-254RX by site staff Comparison of i versus iii: the marked TK-254RX %-scale from iii are transformed into the 5-point scale (≥ 90%, ≥75% to <90%, ≥50% to <75%, >0% to <50%, completely detached); then the 5-point scale assessments from i and iii are compared via 5x5-cross tabulations and Spearman rank correlations.
  Comparison of ii versus iii: the marked TK-254RX %-scale from ii and iii are transformed into the 5-point scale (≥ 90%, ≥75% to <90%, ≥50% to <75%, >0% to <50%, completely detached); then the 5-point scale assessments from ii and iii are compared via 5x5-cross tabulations and Spearman rank correlations.
Characterization of local tolerability during treatment | within 5 minutes after removal of each patch
  The skin will be visually checked and palpated for skin irritation or sensitization by trained personnel.
  Local tolerability will be assessed by the Investigator according to FDA recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Nishiyama, Study Chair — Teikoku Seiyaku Co., Ltd.
Locations (4):
- Germany (4):
  - Medical Practice Ebert, Brühl
  - Medical practice Pabst, Fürstenfeldbruck
  - Medical practice Gastl, Gilching
  - Medical Pracitice Schaale/Bücheler, Rheinbach

IPD SHARING:
Plan to Share IPD: No